CLINICAL TRIAL: NCT04103086
Title: ARomatherapy for Cognitive Trajectory in Chinese After Percutaneous Coronary Intervention (ARCTIC-PCI): a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: ARomatherapy for Cognitive Trajectory in Chinese After Percutaneous Coronary Intervention (ARCTIC-PCI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Wei Yongxiang, Director of Beijing Anzhen Hospital, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BeijingAnzhen-2019-06-PCI
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Percutaneous Coronary Intervention; Aromatherapy; Cognitive function; Randomized Controlled Trial
MeSH Terms: interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: Randomized (two arms), double-blind, placebo-controlled intervention is proposed in this study. 660 participants undergoing PCI are anticipated to be enrolled from the Beijing Anzhen Hospital. Before hospital discharge, participants will be randomly assigned to receive aromatherapy (70% menthol and 30% propanediol) or placebo (10% menthol and 90% propanediol) after PCI for 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, physicians, and outcomes assessors will be blinded to treatment allocation. The sticks of aromatherapy and placebo are the same, and the smell of them is similar. In order to achieve allocation concealment, a web-based central system will automatically assign a random code for each participant. Each bottle of medicine or placebo will be labeled according to the pre-determined random code by an independent agency that does not involve any persons associated with the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The aromatherapy arm (Experimental): Free aromatherapy (70% menthol and 30% propanediol). All participants will receive the standard inhalation method training before hospital discharge.
  The aromatherapy will be given twice daily, one treatment in the morning and one in the evening. At each treatment, 4 deep steady inhalations will be performed, and 10 seconds per inhalation is optimal.
  Interventions: Drug: Aromatherapy
- The placebo arm (Placebo Comparator): Free placebo (10% menthol and 90% propanediol) will be provided for 6 months. The specific method is the same as aromatherapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aromatherapy — Free aromatherapy (70% menthol and 30% propanediol) will be provided for 6 months. All participants will receive the standard inhalation method training before hospital discharge.
  The aromatherapy will be given twice daily, one treatment in the morning and one in the evening. At each treatment, 4 deep steady inhalations will be performed, and 10 seconds per inhalation is optimal.
  Arms: The aromatherapy arm
Drug: Placebo — Free placebo (10% menthol and 90% propanediol) will be provided for 6 months. The specific method is the same as aromatherapy
  Arms: The placebo arm

SUMMARY:
The ARCTIC-PCI (Aromatherapy for Cognitive Trajectory in Chinese after Percutaneous Coronary Intervention) trial is a randomized, double-blind, 2-arm, parallel group, placebo-controlled study to evaluated the effects of aromatherapy in improving cognitive function in post-percutaneous coronary intervention (PCI) patients. The study will recruit 660 patients who undergo a PCI at the Department of Cardiology in Beijing Anzhen Hospital.

Baseline information will be collected prior to PCI, all eligible participants undergoing PCI will be randomly assigned in a 1:1 ratio before hospital discharge to receive aromatherapy (70% menthol and 30% propanediol) or placebo (10% menthol and 90% propanediol). The treatment will last for 6 months in both groups. Cognitive function measurement will be conducted by blinded assessors at baseline (1-3 days before PCI) and at 3- and 6- month after PCI. The primary outcome will be the change in overall cognitive function (MOCA score) from baseline to 6-month after PCI.

DETAILED DESCRIPTION:
The ARCTIC-PCI trial has two objectives. The primary objective is to evaluate the efficacy of aromatherapy (70% menthol and 30% propanediol) in improving cognitive functions in Chinese post-PCI patients. The secondary objective is to evaluate the safety of aromatherapy. We hypothesize that the aromatherapy will result in improved 6- month cognitive functions compared to the placebo (10% menthol and 90% propanediol) among patients accepted a PCI.

Patient recruitment:

The study will be conducted at Beijing Anzhen Hospital. All eligible patients plan to undergo their PCI will be screened for eligibility, written informed consent need to be provided. For patients who meet all inclusion and exclusion criteria, baseline assessment will be carried out 1 to 3 days prior to the PCI.

Randomization and allocation concealment:

Randomization will be conducted after PCI and before hospital discharge. To ensure concealment of the treatment allocation, randomization will be performed by a web-based IT system. All eligible participants will be randomly assigned in a 1:1 ratio to receive aromatherapy (70% menthol and 30% propanediol) or placebo (10% menthol and 90% propanediol). Each sniffin' stick of aromatherapy or placebo will be labeled according to the pre-determined random code by an independent agency that does not involve any persons associated with the trial.

Masking:

Participants, investigators, physicians, and outcomes assessors will be blinded to treatment allocation. The sticks of aromatherapy and placebo are the same, and the smell of them is similar.

Interventions:

Intervention will last for 6 months. All participants will receive the standard inhalation method training before hospital discharge. For both arms, the aromatherapy/placebo will be given twice daily (morning and evening), each time training for 4 times with deep inhalation for 10 seconds.

Supervisory management will be carried out through WeChat app, each day all participants will receive reminders via WeChat through the "group assistant". By the end of the intervention, we will collect all the rest of the medications (menthol/placebo) and the total amount of the rest medication will be assessed to evaluate patients' adherence.

Measurement:

Baseline measurement including the following aspects:

1. Laboratory data including: myocardial enzyme, fasting blood glucose, glycosylated hemoglobin, total cholesterol, low-density cholesterol, high-density cholesterol, triglyceride, high-sensitivity c-reactive protein, creatinine, uric acid, liver function indicators, etc.
2. Genetic testing: APOE genotype.
3. Physical examination: height, weight, blood pressure, heart rate.
4. Clinical data including: left ventricular ejection fraction, heart failure classification, GRACE score, shock, thrombolytic therapy, myocardial infarction classification, type of MI (ST elevation or non-ST elevation), vascular stenosis, coronary artery calcification score, etc.
5. Assessment of olfactory function: collection of prior history of dysosmia or using Sniffin' Sticks test to assess olfactory function.
6. Assessment of cognitive function: The Chinese version of the Montreal Cognitive Assessment (MoCA) will be used, which is translated from the original English version and has been reviewed and authorized by the author of the original edition (Dr. Ziad Nasreddine). The Chinese version of MoCA has been verified in the elderly population in China, with good reliability and validity in screening for MCI and Alzheimer's disease. In addition, we will use internationally recognized scales to evaluate memory, executive function and orientation. All researchers involved in the cognitive function assessment are from the clinical research institute of Peking University, independent of the study sponsor. All cognitive assessors have received MoCA training and obtained official certification.
7. Assessment of depression symptom: The Center for Epidemiologic Studies Depression Scale (CES-D) will be used to measure depression symptoms severity.
8. Surgery information: methods of anesthesia, anesthetic drugs and dosage, duration of PCI, stent type, number of stents, etc.
9. Other information: length of stay in ICU, length of stay in general ward, discharge medications.

Follow-up Assessment： All participants will be invited back to hospital twice at 3- and 6- month after PCI. Cognitive functions will be assessed by the same assessors using the same methods as baseline.

Adverse events:

During the 6-month follow-up period will be recorded, which are defined as any of the unexpected signs (such as abnormal lab values), symptoms, or diseases, whether or not associated with aromatherapy.

Study-related adverse reactions including 1) respiratory allergy and 2) sneeze. Severe adverse events (SAE) during follow-up are defined as any of the following:1) all-cause mortality, 2) hospitalization for cardiovascular disease, 3) re-myocardial infarction and 4) stroke.

Sample Size Calculation:

The total number of subjects required for this study is 330:330 patients per group. This number was determined on the basis of the following hypotheses, with reference obtained from the FINGER trial (Lancet 2015;385:2255-2263), Xie et.al (JACC 2019;73: 3041-3050) and other related observational studies.

1. A decrease of 0.2 Z-score with a standard deviation of 0.3 at 6-month post-PCI in the control group
2. Intervention will reduce the overall cognitive decline by 40%, that is a decrease of 0.12 Z-score at 6-month post-PCI in the intervention group.
3. α risk of 5% and β risk of 10%
4. the maximum lost to follow-up rate:10%

Statistical Analysis:

The principal analysis will be a modified intention-to-treat (ITT) analysis on patients with at least one follow-up included in the study. The primary and continuous secondary outcomes are repeated measures, and linear mixed models will be used for analysis. All continuous outcomes will be standardized according to the mean and standard deviation of their baseline values, and z-score of each variable will be obtained. Modified Poisson regression analysis will be used for binary secondary outcomes.

Sensitivity analyses include: 1) ITT analysis including all participants, with missing data being imputed by using multiple imputation method. 2) Only include patients with both follow-up measurements. 3) For the primary outcome, we will also test if the intervention effect is modified by baseline characteristics.

Statistical analyses will be carried out using the SAS Enterprise Guide 7.13 (SAS Institute Inc, Cary, NC)

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 50 and 75 years old.
2. Patients with unstable angina, ST-segment elevation or non-ST elevation myocardial infarction who need stent implantation.
3. Willing to come to hospital at 3- and 6- month after PCI.
4. Signed informed consent.

Exclusion Criteria:

1. Emergency patients.
2. Prior history of CABG(Coronary Artery Bypass Grafting),or other cardiac surgery.
3. Prior history of heart failure.
4. Prior history of atrial fibrillation.
5. Prior history of allergic rhinitis, sinusitis, asthma and COPD.
6. Deafness, mental illness including severe depression, and inability to communicate properly.
7. Prior history of stroke.
8. Prior history of brain tumor, traumatic brain injury, or other brain surgery.
9. Relatives of researcher or management personnel.
10. Family members been enrolled in the study.
11. Known mild cognitive impairment or dementia.
12. Mild cognitive impairment and dementia identified by cognitive function assessment before PCI.
13. Prior history of smell disorder or decreased/loss of olfactory functions assessed by the Sniffin' Sticks test.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the overall cognitive function at 6 months after PCI | before and after 6-month intervention
  Changes in the overall cognitive function in the Aromatherapy group versus changes in the overall cognitive function in the placebo group. MOCA (MOCA-Montreal Cognitive Assessment) will be used to measure the overall cognitive function.
Changes in the overall cognitive function at 3 months after PCI | before and after 6-month intervention
  Changes in the overall cognitive function in the Aromatherapy group versus changes in the overall cognitive function in the placebo group. MOCA (MOCA-Montreal Cognitive Assessment) will be used to measure the overall cognitive function.
Changes in the memory function at 3- and 6- month after PCI | before and after 3- and 6-month intervention
  Changes in the memory function in the Aromatherapy group versus changes in the memory function in the placebo group. The test of Word-List Immediate and Delayed Recall will be used to access the memory.
Changes in the executive function: semantic fluency, at 3- and 6- month after PCI | before and after 3- and 6-month intervention
  Changes in the executive function of semantic fluency in the Aromatherapy group versus changes in the executive function in the placebo group. Animal Fluency Test will be used to access participants' semantic fluency.
Changes in the executive function: visual attention, at 3- and 6- month after PCI | before and after 3- and 6-month intervention
  Changes in the executive function of visual attention in the Aromatherapy group versus changes in the executive function in the placebo group. Chinese version of Trails Making Test will be used to access patients' visual attention.
Changes in the orientation function at 3- and 6- month after PCI | before and after 3- and 6-month intervention
  Changes in the orientation function in the Aromatherapy group versus changes in the orientation function in the placebo group. MoCA Orientation function test will be used to access the orientation function.
The proportion of patients with mild cognitive impairment at 3- and 6- month after PCI | before and after 3- and 6- month intervention
  The proportion of patients with mild cognitive impairment in the Aromatherapy group versus the proportion of patients with mild cognitive impairment in the placebo group.
  Mild cognitive impairment is measured by using different cut-off points for cognitive function scores in the Chinese version of MOCA. For participants with low, secondary, and high education levels, mild cognitive impairment is defined as having an overall cognitive function score <19, <22, and <24 respectively. Low education level, secondary education level and high education level are defined as the number of years of education ≤6 years, 7-12 years and > 12 years respectively.

IPD SHARING:
Plan to Share IPD: Undecided
All data of this trial can be obtained on request.

REFERENCES:
- [Background] Xie W, Zheng F, Yan L, Zhong B. Cognitive Decline Before and After Incident Coronary Events. J Am Coll Cardiol. 2019 Jun 25;73(24):3041-3050. doi: 10.1016/j.jacc.2019.04.019. PMID 31221251